CLINICAL TRIAL: NCT03043456
Title: Evaluation of Patient Satisfaction and Microbiological Changes in Injectable Thermoplastic Resin and Conventional Acrylic Resin Complete Dentures
Brief Title: Patient Satisfaction and Microbial Changes in Complete Dentures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdel Hamid, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 28806032102395
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Satisfaction; Microbial Colonization
MeSH Terms: conditions — Personal Satisfaction; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: prospective , parallel, randomized clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be blinded regarding the statistician who is responsible for data analysis.
  The participant patients will be blinded. The outcome assessor for patient satisfaction can be blinded during the questionnaire. On the other hand, Microbial count assessor will not be blinded during swab taking while the lab technician can be blinded. but The operator cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermoplastic Resin group (Active Comparator): Thermoplastic complete denture placement is done (Thermoplastic Comfort Systems, inc.)
  Interventions: Device: Thermoplastic complete denture
- conventional acrylic resin group (Placebo Comparator): Conventional acrylic resin complete denture placement is done. (Acrostone, inc.)
  Interventions: Device: Conventional acrylic resin complete denture

INTERVENTIONS:
Device: Thermoplastic complete denture — A device used to substitute the teeth for edentulous patients made of thermoplastic resin
  Arms: Thermoplastic Resin group
Device: Conventional acrylic resin complete denture — A device used to substitute the teeth for edentulous patients made of acrylic resin
  Arms: conventional acrylic resin group

SUMMARY:
In this research, the investigators are comparing the new thermoplastic material side by side with the conventional poly methyl methacrylate for fully edentulous patients measuring their satisfaction and microbiological count.

DETAILED DESCRIPTION:
The restoration of masticatory function and aesthetics is an important aim in dentistry mainly when patients present with extensive tooth loss. The loss of tooth in elderly patients not only impairs the stomatognathic system but also their psychological status and quality of life.so an important criteria's for the success of dentures are patient's expectations and the ability of the denture to replace the lost masticatory efficiency.

The acrylic resin was first used in 1936; it was in that time the best alternative for vulcanized rubber. Where it is characterized by superior characteristics and became the most popular material used since then. Nonetheless, it has some problems such as polymerization shrinkage, weak flexural, lower impact strength, and low fatigue resistance. These often lead to denture failure during chewing or when fall out of the patient's hand. In order to enhance some properties of PMMA, various efforts have been taken including addition of metal wires or plates, fibers, metal inserts, and modification of chemical structure. In recent years, nylon polymer has attracted attention as a denture base material.

Thermoplastic nylon like materials or polyamides were introduced and first used in dentistry in 1950. The polyamide are uniquely characterized by high esthetics especially in removable partial dentures, where retentive components are recommended anteriorly by this material which provide high elasticity we can make the retentive components using the same material and eliminate the metallic clasps.

Polyamides are characterized by low weight and flexibility make it more patient satisfactory and fortunately it has no monomer remnants that may affect patient health and causes allergy. Thermoplastic polyamides have almost no porosity which eliminates water sorption. The technique used for its fabrication is injection molding technique which is more dimension accurate than packing mold technique.

Valplast was initially used just over 50 years ago and has been used in modern dentistry since the mid-fifties. A variation of nylon, which is far more flexible and stronger than poly methyl methacrylate resin, is used in many alternative partial dentures. Valplast flexible dentures are used for full sets of dentures especially in cases of acrylic allergy which represent 20% of the population.

Comparative Evaluation of Impact and Flexural Strength is done to four types of Four Commercially Available Flexible Denture Base Materials. Valplast had the maximum impact strength, so these materials should be used in less undercut areas for long-term interim removable partial dentures.

A study done by investigators who evaluated the surface roughness of four thermoplastic (polyamide: Valplast, Lucitone FRS, polyethylene terephthalate: EstheShot, and polyester: EstheShot Bright) and two conventional acrylic (Heat-polymerizing: Urban, and Pour type auto-polymerizing: Pro-Cast DSP) denture bases by using scratch test. The results showed that the surface of thermoplastic denture base resins was easily damaged compared with polymethyl methacrylate which can cause discomfort to patients and also discoloration.

Complete Dentures Made with High Impact and Flexible Resins were evaluated. There was statistically significant difference for masticatory performance in wet and dry weight values of hard food, but there was no statistically significant difference for masticatory performance in wet and dry weight values of soft food between the conventional and flexible dentures. Though masticatory efficiency and performance were found to be better for patient's dentures made with Polymethyl methacrylate (PMMA), a statistically significant number of patients reported that the flexible dentures were more satisfying than the conventional dentures.

Another study was done to evaluate the patients inflamatory response. patients received acrylic complete denture were associated with significant high levels of proinflammatory salivary cytokines (TNF-α and IL-6) in comparison to their corresponding levels in the thermoplastic polyamide complete denture patients. The high levels of pro-inflammatory salivary cytokines (TNF-α and IL-6) that were found in saliva of control group patients may be linked to their protective effect against tissue inflammation caused by release of residual monomer.

Adherence of Candida albicans to Flexible Denture Base Material was studied and concluded C. albicans has lesser opportunities to adhere on flexible denture than on acrylic resin denture base materials.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous
* No bone irregularities, no bone specules, mild to moderate undercut.
* Good oral hygiene
* Should be co-operative
* No serious systemic disease
* No TMJ Problems

Exclusion Criteria:

* Bone irregularities , soft tissue ulcerations , severe undercuts
* Serious systemic problem
* Patient with xerostomia
* Severely resorbed ridge
* Logistic or physical reasons that could affect follow-up,
* Psychiatric problems
* Medically compromised patients & those with neuromascular disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Patient satisfaction | 0 months , 3 months , 6 months
  Questionnaire

SECONDARY OUTCOMES:
changes in Microbial count | 0 months , 3 months , 6 months
  CFU

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Rekaby, Ph.D., Study Chair — Cairo University; Azza A Farahat, Ph.D., Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No
Data will be available through contact by email of the principle investigator. (gazar_fantasy@yahoo.com)

REFERENCES:
- [Background] Singh K, Aeran H, Kumar N, Gupta N. Flexible thermoplastic denture base materials for aesthetical removable partial denture framework. J Clin Diagn Res. 2013 Oct;7(10):2372-3. doi: 10.7860/JCDR/2013/5020.3527. Epub 2013 Oct 5. PMID 24298532
- [Background] Osada H, Shimpo H, Hayakawa T, Ohkubo C. Influence of thickness and undercut of thermoplastic resin clasps on retentive force. Dent Mater J. 2013;32(3):381-9. doi: 10.4012/dmj.2012-284. PMID 23718997
- [Background] Goiato MC, Santos DM, Haddad MF, Pesqueira AA. Effect of accelerated aging on the microhardness and color stability of flexible resins for dentures. Braz Oral Res. 2010 Jan-Mar;24(1):114-9. doi: 10.1590/s1806-83242010000100019. PMID 20339724
- [Background] Samet N, Tau S, Findler M, Susarla SM, Findler M. Flexible, removable partial denture for a patient with systemic sclerosis (scleroderma) and microstomia: a clinical report and a three-year follow-up. Gen Dent. 2007 Nov-Dec;55(6):548-51. PMID 18050582
- [Background] León BL, Del Bel Cury AA, Rodrigues Garcia RC. Loss of residual monomer from resilient lining materials processed by different methods. Rev Odontol Ciêc. 2008;23:215-9.
- [Background] Bayraktar G, Guvener B, Bural C, Uresin Y. Influence of polymerization method, curing process, and length of time of storage in water on the residual methyl methacrylate content in dental acrylic resins. J Biomed Mater Res B Appl Biomater. 2006 Feb;76(2):340-5. doi: 10.1002/jbm.b.30377. PMID 16161124
- [Background] Urban VM, Machado AL, Vergani CE, Giampaolo ET, Pavarina AC, de Almeida FG, Cass QB. Effect of water-bath post-polymerization on the mechanical properties, degree of conversion, and leaching of residual compounds of hard chairside reline resins. Dent Mater. 2009 May;25(5):662-71. doi: 10.1016/j.dental.2008.10.017. Epub 2009 Jan 10. PMID 19135715
- [Background] NIRONEN P. Some possible uses for acrylic resins in dentistry. Odontol Tidskr. 1950;58(2):118-25. No abstract available. PMID 14785900
- [Background] Giunta JL, Grauer I, Zablotsky N. Allergic contact stomatitis caused by acrylic resin. J Prosthet Dent. 1979 Aug;42(2):188-90. doi: 10.1016/0022-3913(79)90173-2. No abstract available. PMID 287797
- [Background] Weaver RE, Goebel WM. Reactions to acrylic resin dental prostheses. J Prosthet Dent. 1980 Feb;43(2):138-42. doi: 10.1016/0022-3913(80)90176-6. PMID 6985962